CLINICAL TRIAL: NCT06828718
Title: Comparison of the Prognosis and Safety of Different Neoadjuvant Treatment Modalities in Patients With Locally Advanced Esophageal Squamous Cell Carcinoma: A National Multicenter Real-World Study(NEO-EC）
Brief Title: The Neoadjuvant Treatment Modalities in Patients With Locally Advanced Esophageal Squamous Cell Carcinoma (NEO-EC）
Acronym: NEO-EC
Status: Active, not recruiting | Type: Observational
Sponsor: Hebei Medical University Fourth Hospital (Other)
Collaborators: Tianjin Medical University Cancer Institute and Hospital (Other); Fujian Cancer Hospital (Other Government); Shandong Cancer Hospital and Institute (Other); Shanxi Province Cancer Hospital (Other); Jiangsu Cancer Institute & Hospital (Other); Sichuan Cancer Hospital and Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 2025KS008
Record Dates: First submitted 2025-02-10; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Esophageal Carcinoma
Keywords: Esophageal Carcinoma; Neoadjuvant therapy; Prognosis
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Neoadjuvant chemoradiotherapy: Patients with locally advanced esophageal squamous cell carcinoma received neoadjuvant chemoradiotherapy and then underwent surgical resection
- Neoadjuvant chemotherapy: Patients with locally advanced esophageal squamous cell carcinoma received neoadjuvant chemotherapy followed by surgical resection
- Neoadjuvant chemotherapy combined with immunotherapy: Patients with locally advanced esophageal squamous cell carcinoma underwent surgical resection after neoadjuvant chemotherapy combined with immunotherapy
- Neoadjuvant chemoradiotherapy combined with immunotherapy: Patients with locally advanced esophageal squamous cell carcinoma underwent surgical resection after neoadjuvant chemoradiotherapy combined with immunotherapy

SUMMARY:
The prognosis and safety of patients with locally advanced esophageal squamous cell carcinoma were compared with different neoadjuvant therapy modes in multi-cancer centers in China

DETAILED DESCRIPTION:
Neoadjuvant chemoradiotherapy or neoadjuvant chemotherapy combined with surgery are the main treatment methods for patients with locally advanced esophageal squamous cell carcinoma, but some patients still have local recurrence or distant metastasis after surgery. In the era of immunotherapy, immune checkpoint inhibitor monotherapy or combined chemotherapy has become the first-line and second-line standard treatment for recurrent or metastatic esophageal cancer and has been recommended by NCCN guidelines. However, relevant studies on immunotherapy's participation in neoadjuvant therapy have shown good results, but it is still in its initial stage, and its efficacy needs further research and discussion.Thus, we compared the prognosis and safety of patients with locally advanced esophageal squamous cell carcinoma who received different neoadjuvant therapy before surgery, including neoadjuvant chemoradiotherapy, neoadjuvant chemotherapy, neoadjuvant chemotherapy combined with immunotherapy, and neoadjuvant chemoradiotherapy combined with immunotherapy in several cancer centers in China.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years, male or female;
2. KPS score (KPS) ≥70;
3. Esophageal squamous cell carcinoma confirmed by histopathology;
4. Clinical stage cT1b-4aN+M0,T3-4aN0M0;
5. Surgical resection was performed after 2~4 cycles of neoadjuvant therapy.
6. Expected survival > 6 months.

Exclusion Criteria:

1. Have a history of other malignancies (except for cancer in situ that has been cured and other malignancies that have been cured for more than 5 years);
2. There are contraindications of immunotherapy or chemoradiotherapy;
3. Inability to tolerate or refuse surgery;
4. Distant metastasis has occurred;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: we compared the prognosis and safety of patients with locally advanced esophageal squamous cell carcinoma who received different neoadjuvant therapy before surgery, including neoadjuvant chemoradiotherapy, neoadjuvant chemotherapy, neoadjuvant chemotherapy combined with immunotherapy, and neoadjuvant chemoradiotherapy combined with immunotherapy in several cancer centers in China.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of pathological complete response rate (pCR) after surgical resection in patients with locally advanced esophageal squamous cell carcinoma receiving different neoadjuvant therapy | 2015.1.1-2023.12.31
  Pathological complete response (pCR) is defined as the absence of residual tumor cells after evaluation of removed tumor tissue and regional lymph nodes.
Comparison of major pathological response (MPR) after surgical resection in patients with locally advanced esophageal squamous cell carcinoma receiving different neoadjuvant therapy | 2015.1.1-2023.12.31
  Major pathological response (MPR) is defined as a tumor that has significantly shrunk or decreased in the pathological evaluation, but still has a small number of residual tumor cells.

SECONDARY OUTCOMES:
Comparison of the overall survival (OS) after surgical resection in patients with locally advanced esophageal squamous cell carcinoma receiving different neoadjuvant therapy | 2015.1.1-2025.12.31
  OS is defined as the time from the start of enrollment to death from any cause
Comparison of the disease-free survival (DFS) after surgical resection in patients with locally advanced esophageal squamous cell carcinoma receiving different neoadjuvant therapy | 2015.1.1-2025.12.31
  DFS difined as the time between the start of the enrollment and the recurrence of disease, or death from any cause.

OTHER OUTCOMES:
Comparison of incidence of treatment-related adverse evants after surgical resection in patients with locally advanced esophageal squamous cell carcinoma receiving different neoadjuvant therapy | 2015.1.1-2025.12.31
  Adverse events are observed during the course of the study and assessed according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI CTCAE V5.0).

CONTACTS AND LOCATIONS:
Locations (1):
- Shijiazhuang, Hebei, China